CLINICAL TRIAL: NCT05592951
Title: Randomized Trial to Assess the Safety and Tolerability of a Novel Amino-acid Based Hydration Drink in Healthy Volunteers
Brief Title: Safety and Tolerability of a Novel Amino-acid Based Hydration Drink in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO-FY2023-5
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Safety; Tolerance
Keywords: Liquid IV; amino acids; electrolytes
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo once daily (Placebo Comparator): 1 stick pack dissolved in water once daily prior to breakfast
  Interventions: Dietary Supplement: Crystal Light (once serving)
- Test beverage once daily (Experimental): 1 stick pack dissolved in water once daily prior to breakfast
  Interventions: Dietary Supplement: Liquid IV with amino acids (one serving)
- Test beverage twice daily (Experimental): 2 stick packs dissolved in water, one packet at a time twice daily (after lunch and after dinner)
  Interventions: Dietary Supplement: Liquid IV with amino acids (two servings)
- Test beverage three times daily (Experimental): 3 stick packs dissolved in water, one packet at a time three times daily (after breakfast, lunch, and dinner)
  Interventions: Dietary Supplement: Liquid IV with amino acids (three servings)

INTERVENTIONS:
Dietary Supplement: Crystal Light (once serving) — Citric Acid, Potassium Citrate, Sodium Citrate, Aspartame (Phenylketonurics: Contains Phenylalanine), Magnesium Oxide, Maltodextrin, Contains Less than 2% of Natural Flavor, Acesulfame Potassium, Soy Lecithin, Yellow 5, Artificial Color.
  Arms: Placebo once daily
Dietary Supplement: Liquid IV with amino acids (one serving) — Allulose, L-Alanine, L-Glutamine, Citric Acid, Sodium chloride, Lemon Lime Flavorings, Potassium Citrate, Trisodium Citrate Dihydrate, Dipotassium Phosphate, Syloid Silicon Dioxide, Stevia, Vitamin C, Vitamin B3, Calcium Pantothenate B5 (Vitamin B5), Vitamin B6, Vitamin B12. Liquid IV packets contain: sodium and potassium.
  Arms: Test beverage once daily
Dietary Supplement: Liquid IV with amino acids (two servings) — Allulose, L-Alanine, L-Glutamine, Citric Acid, Sodium chloride, Lemon Lime Flavorings, Potassium Citrate, Trisodium Citrate Dihydrate, Dipotassium Phosphate, Syloid Silicon Dioxide, Stevia, Vitamin C, Vitamin B3, Calcium Pantothenate B5 (Vitamin B5), Vitamin B6, Vitamin B12. Liquid IV packets contain: sodium and potassium.
  Arms: Test beverage twice daily
Dietary Supplement: Liquid IV with amino acids (three servings) — Allulose, L-Alanine, L-Glutamine, Citric Acid, Sodium chloride, Lemon Lime Flavorings, Potassium Citrate, Trisodium Citrate Dihydrate, Dipotassium Phosphate, Syloid Silicon Dioxide, Stevia, Vitamin C, Vitamin B3, Calcium Pantothenate B5 (Vitamin B5), Vitamin B6, Vitamin B12. Liquid IV packets contain: sodium and potassium.
  Arms: Test beverage three times daily

SUMMARY:
The nutrient composition of this product is similar to the existing Liquid IV "hydration multiplier" product already on the market but with the addition of amino acids. With such low quantities of amino acids, in particular as compared to the amounts consumed in normal diets, there is no reason to believe that the product would cause any adverse outcomes. However, since no research has been done on the safety of regular consumption of this product, this study will evaluate the safety of the product with regards to routing blood chemistries and other variables. Specifically, standard testing will be performed including a measurement of vital signs, comprehensive metabolic panel, hematology panel, urinalysis, and quantification of triiodothyronine, thyroxine, and thyroid stimulating hormone. A questionnaire will also be used to assess product tolerability.

DETAILED DESCRIPTION:
Maintaining adequate hydration is essential to optimal health, as well as athletic performance. When individuals exercise (in particular in a warm environment), they can lose excessive amounts of fluids along with necessary electrolytes (e.g., sodium, potassium, chloride) through sweating. With dehydration, individuals may feel sluggish and can experience impaired physical performance.

The use of electrolytes (sodium in particular) has been used for decades to aid athlete hydration and has led to the development of various sport drinks (e.g., Gatorade, Powerade) -which also include small amounts of carbohydrate. The addition of amino acids to electrolyte solutions has previously been demonstrated to further increase the transport of water and sodium from the jejunum (small intestine). Separate research also showed an amino acid and electrolyte drink increased cellular hydration compared to flavored water and electrolyte only drinks. A 2019 study found that amino acids hydration increased beverage hydration index (BHI)-a measure of fluid balance following consumption of a beverage and was age dependent.

Amino acids supplementation has been popular for some time among athletes due to other potential performance benefits including changes to anabolic hormone levels, alterations to energy consumption, and mental endurance. Further, amino acids may reduce post-exercise muscle soreness and aid in recovery.

The electrolyte amino-acid test product is a powder provided in individual stick packs and contains L-Alanine and L-Glutamine as well as 5 essential vitamins including Vitamins B3, B5, B6, B12 and Vitamin C. It is gluten-, soy-, and dairy-free, and provides electrolytes well below the daily value. The daily value (DV) tells us how much a particular nutrient in a serving of a food product contributes to a daily diet, based on a standard 2000 calorie diet. Despite what the name suggests, this product is taken orally, not intravenously. Liquid IV packets contain: sodium (510 mg, 22%DV) and potassium (380 mg, 8%DV). These packets contain a small percentage of the needed total electrolytes but adequate amounts to replace lost electrolytes as a result of physical activity.

The nutrient composition of this product is similar to the existing Liquid IV "hydration multiplier" product already on the market but with the addition of amino acids. With such low quantities of amino acids, in particular as compared to the amounts consumed in normal diets, there is no reason to believe that the product would cause any adverse outcomes. However, since no research has been done on the safety of regular consumption of this product, this study will evaluate the safety of the product with regards to routing blood chemistries and other variables. Specifically, standard testing will be performed including a measurement of vital signs, comprehensive metabolic panel, hematology panel, urinalysis, and quantification of triiodothyronine, thyroxine, and thyroid stimulating hormone. A questionnaire will also be used to assess product tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18-29.9 kg/m2
* able to fast overnight

Exclusion Criteria:

* tobacco user
* history of heart disease/cardiovascular disease
* hypertensive (140/90 mmHg or less)
* diabetes
* history of immune disorder
* history of kidney disease
* hepatic impairment or disease
* history of unstable thyroid
* abnormality or obstruction of the gastrointestinal tract precluding swallowing
* abnormal digestion conditions
* previously diagnosed major affective disorder
* psychiatric disorder that required hospitalization in prior year
* history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening)
* no known sensitivity or allergy to any of the study products
* consumption of alcohol-containing beverages within 24 hours of testing
* consumption of caffeine-containing beverages within 24 hours of testing
* active infection or illness of any kind
* if female, lactating, pregnant, or planning to become pregnant during the study
* receipt or use of an investigational product in another research study or change in medication, dietary supplementation, or significant change in diet/exercise regimen within 28 days prior to baseline/visit 2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Alanine transaminase | baseline
  Alanine transaminase measured as part of metabolic panel with units IU/L
Alanine transaminase | 2 weeks of assigned treatment
  Alanine transaminase measured as part of metabolic panel with units IU/L
Alanine transaminase | 4 weeks of assigned treatment
  Alanine transaminase measured as part of metabolic panel with units IU/L
Aspartate transferase | baseline
  Aspartate transferase measured as part of comprehensive metabolic panel with units IU/L
Aspartate transferase | 2 weeks of assigned treatment
  Aspartate transferase measured as part of comprehensive metabolic panel with units IU/L
Aspartate transferase | 4 weeks of assigned treatment
  Aspartate transferase measured as part of comprehensive metabolic panel with units IU/L
Albumin | baseline
  Albumin measured as part of comprehensive metabolic panel with units g/dL
Albumin | 2 weeks of assigned treatment
  Albumin measured as part of comprehensive metabolic panel with units g/dL
Albumin | 4 weeks of assigned treatment
  Albumin measured as part of comprehensive metabolic panel with units g/dL
Alkaline phosphatase | baseline
  Alkaline phosphatase measured as part of comprehensive metabolic panel with units IU/L
Alkaline phosphatase | 2 weeks of assigned treatment
  Alkaline phosphatase measured as part of comprehensive metabolic panel with units IU/L
Alkaline phosphatase | 4 weeks of assigned treatment
  Alkaline phosphatase measured as part of comprehensive metabolic panel with units IU/L
total bilirubin | baseline
  total bilirubin measured as part of comprehensive metabolic panel with units mg/dL
total bilirubin | 2 weeks of assigned treatment
  total bilirubin measured as part of comprehensive metabolic panel with units mg/dL
total bilirubin | 4 weeks of assigned treatment
  total bilirubin measured as part of comprehensive metabolic panel with units mg/dL
blood urea nitrogen mg/dL | baseline
  blood urea nitrogen as part of comprehensive metabolic panel with unite
blood urea nitrogen | 2 weeks of assigned treatment
  blood urea nitrogen as part of comprehensive metabolic panel with units mg/dL
blood urea nitrogen | 4 weeks of assigned treatment
  blood urea nitrogen as part of comprehensive metabolic panel with units mg/dL
calcium | baseline
  calcium as part of comprehensive metabolic panel with units mg/dL
calcium | 2 weeks of assigned treatment
  calcium as part of comprehensive metabolic panel with units mg/dL
calcium | 4 weeks of assigned treatment
  calcium as part of comprehensive metabolic panel with units mg/dL
carbon dioxide | baseline
  carbon dioxide as part of comprehensive metabolic panel with units mmol/L
carbon dioxide | 2 weeks of assigned treatment
  carbon dioxide as part of comprehensive metabolic panel with units mmol/L
carbon dioxide | 4 weeks of assigned treatment
  carbon dioxide as part of comprehensive metabolic panel with units mmol/L
chloride | baseline
  chloride as part of comprehensive metabolic panel with units mmol/L
chloride | 2 weeks of assigned treatment
  chloride as part of comprehensive metabolic panel with units mmol/L
chloride | 4 weeks of assigned treatment
  chloride as part of comprehensive metabolic panel with units mmol/L
creatinine | baseline
  creatinine as part of comprehensive metabolic panel with units mg/dL
creatinine | 2 weeks of assigned treatment
  creatinine as part of comprehensive metabolic panel with units mg/dL
creatinine | 4 weeks of assigned treatment
  creatinine as part of comprehensive metabolic panel with units mg/dL
estimated glomerular filtration rate calculation | baseline
  estimated glomerular filtration rate calculation as part of comprehensive metabolic panel with units mL/min/1.73
estimated glomerular filtration rate calculation | 2 weeks of assigned treatment
  estimated glomerular filtration rate calculation as part of comprehensive metabolic panel with units mL/min/1.73
estimated glomerular filtration rate calculation | 4 weeks of assigned treatment
  estimated glomerular filtration rate calculation as part of comprehensive metabolic panel with units mL/min/1.73
blood glucose | baseline
  glucose as part of comprehensive metabolic panel with units mg/dL
blood glucose | 2 weeks of assigned treatment
  glucose as part of comprehensive metabolic panel with units mg/dL
blood glucose | 4 weeks of assigned treatment
  glucose as part of comprehensive metabolic panel with units mg/dL
potassium | baseline
  potassium as part of comprehensive metabolic panel with units mmol/L
potassium | 2 weeks of assigned treatment
  potassium as part of comprehensive metabolic panel with units mmol/L
potassium | 4 weeks of assigned treatment
  potassium as part of comprehensive metabolic panel with units mmol/L
total protein as part of comprehensive metabolic panel with units g/dL | baseline
  total protein
total protein as part of comprehensive metabolic panel with units g/dL | 2 weeks of assigned treatment
  total protein
total protein as part of comprehensive metabolic panel with units g/dL | 4 weeks of assigned treatment
  total protein
sodium | baseline
  sodium as part of comprehensive metabolic panel with units mmol/L
sodium | 2 weeks of assigned treatment
  sodium as part of comprehensive metabolic panel with units mmol/L
sodium | 4 weeks of assigned treatment
  sodium as part of comprehensive metabolic panel with units mmol/L
total globulin | baseline
  total globulin as part of comprehensive metabolic panel with units g/dL
total globulin | 2 weeks of assigned treatment
  total globulin as part of comprehensive metabolic panel with units g/dL
total globulin | 4 weeks of assigned treatment
  total globulin as part of comprehensive metabolic panel with units g/dL
albumin/globulin ratio | baseline
  albumin/globulin ratio as part of comprehensive metabolic panel
albumin/globulin ratio | 2 weeks of assigned treatment
  albumin/globulin ratio as part of comprehensive metabolic panel
albumin/globulin ratio | 4 weeks of assigned treatment
  albumin/globulin ratio as part of comprehensive metabolic panel
blood urea nitrogen/creatinine ratio | baseline
  blood urea nitrogen/creatinine ratio as part of comprehensive metabolic panel
blood urea nitrogen/creatinine ratio | 2 weeks of assigned treatment
  blood urea nitrogen/creatinine ratio as part of comprehensive metabolic panel
blood urea nitrogen/creatinine ratio | 4 weeks of assigned treatment
  blood urea nitrogen/creatinine ratio as part of comprehensive metabolic panel
Hematocrit | baseline
  Hematocrit as part of complete blood count panel with differential test measured as percentage
Hematocrit | 2 weeks of assigned treatment
  Hematocrit as part of complete blood count panel with differential test measured as percentage
Hematocrit | 4 weeks of assigned treatment
  Hematocrit as part of complete blood count panel with differential test measured as percentage
hemoglobin | baseline
  hemoglobin as part of complete blood count panel with differential test measured as g/dL
hemoglobin | 2 weeks of assigned treatment
  hemoglobin as part of complete blood count panel with differential test measured as g/dL
hemoglobin | 4 weeks of assigned treatment
  hemoglobin as part of complete blood count panel with differential test measured as g/dL
mean corpuscular volume | baseline
  mean corpuscular volume as part of complete blood count panel with differential test measured as femtoliter
mean corpuscular volume | 2 weeks of assigned treatment
  mean corpuscular volume as part of complete blood count panel with differential test measured as femtoliter
mean corpuscular volume | 4 weeks of assigned treatment
  mean corpuscular volume as part of complete blood count panel with differential test measured as femtoliter
mean corpuscular hemoglobin concentration | baseline
  mean corpuscular hemoglobin concentration as part of complete blood count panel with differential test measured as g/dL
mean corpuscular hemoglobin concentration | 2 weeks of assigned treatment
  mean corpuscular hemoglobin concentration as part of complete blood count panel with differential test measured as g/dL
mean corpuscular hemoglobin concentration | 4 weeks of assigned treatment
  mean corpuscular hemoglobin concentration as part of complete blood count panel with differential test measured as g/dL
White blood cell distribution (absolute) | baseline
  absolute measures of white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes per microliter as part of complete blood count panel
White blood cell distribution (absolute) | 2 weeks of assigned treatment
  absolute measures of white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes per microliter as part of complete blood count panel
White blood cell distribution (absolute) | 4 weeks of assigned treatment
  absolute measures of white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes per microliter as part of complete blood count panel
White blood cell distribution (percentage) | baseline
  percentages of white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes out of total white blood cells.
White blood cell distribution (percentage) | 2 weeks of assigned treatment
  percentages of white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes out of total white blood cells.
White blood cell distribution (percentage) | 4 weeks of assigned treatment
  percentages of white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes out of total white blood cells.
Red cell distribution width | baseline
  red cell distribution width as part of complete blood count panel with differential test measured as percentage
Red cell distribution width | 2 weeks of assigned treatment
  red cell distribution width as part of complete blood count panel with differential test measured as percentage
Red cell distribution width | 4 weeks of assigned treatment
  red cell distribution width as part of complete blood count panel with differential test measured as percentage
platelet count | baseline
  platelet count per microliter as part of complete blood count panel with differential test
platelet count | 2 weeks of assigned treatment
  platelet count per microliter as part of complete blood count panel with differential test
platelet count | 4 weeks of assigned treatment
  platelet count per microliter as part of complete blood count panel with differential test
red cell count | baseline
  red cell count per microliter as part of complete blood count panel with differential test
red cell count | 2 weeks of assigned treatment
  red cell count per microliter as part of complete blood count panel with differential test
red cell count | 4 weeks of assigned treatment
  red cell count per microliter as part of complete blood count panel with differential test
white cell count | baseline
  white cell count per microliter as part of complete blood count panel with differential test
white cell count | 2 weeks of assigned treatment
  white cell count per microliter as part of complete blood count panel with differential test
white cell count | 4 weeks of assigned treatment
  white cell count per microliter as part of complete blood count panel with differential test
Triiodothyronine | baseline
  Triiodothyronine measured in blood as ng/dL
Triiodothyronine | 2 weeks of assigned treatment
  Triiodothyronine measured in blood as ng/dL
Triiodothyronine | 4 weeks of assigned treatment
  Triiodothyronine measured in blood as ng/dL
Thyroxine | baseline
  Thyroxine measured in blood as ug/dL
Thyroxine | 2 weeks of assigned treatment
  Thyroxine ug/dL measured in blood as ug/dL
Thyroxine | 4 weeks of assigned treatment
  Thyroxine ug/dL measured in blood as ug/dL
thyroid stimulating hormone | baseline
  Thyroxine measured in blood as micro-IU/dL
thyroid stimulating hormone | 2 weeks of assigned treatment
  Thyroxine measured in blood as micro-IU/dL
thyroid stimulating hormone | 4 weeks of assigned treatment
  Thyroxine measured in blood as micro-IU/dL
Urine Color | baseline
  Urine color as reported in complete urinalysis
Urine Color | 2 weeks of assigned treatment
  Urine color as reported in complete urinalysis
Urine Color | 4 weeks of assigned treatment
  Urine color as reported in complete urinalysis
Urine appearance | baseline
  Urine appearance as reported in complete urinalysis
Urine appearance | 2 weeks of assigned treatment
  Urine appearance as reported in complete urinalysis
Urine appearance | 4 weeks of assigned treatment
  Urine appearance as reported in complete urinalysis
Urine specific gravity | baseline
  Urine specific gravity as reported in complete urinalysis
Urine specific gravity | 2 weeks of assigned treatment
  Urine specific gravity as reported in complete urinalysis
Urine specific gravity | 4 weeks of assigned treatment
  Urine specific gravity as reported in complete urinalysis
Urine potential of hydrogen | baseline
  Urine potential of hydrogen (pH) as reported in complete urinalysis
Urine potential of hydrogen | 2 weeks of assigned treatment
  Urine potential of hydrogen (pH) as reported in complete urinalysis
Urine potential of hydrogen | 4 weeks of assigned treatment
  Urine potential of hydrogen (pH) as reported in complete urinalysis
Protein in urine | baseline
  Protein, if present, measured in urine in complete urinalysis
Protein in urine | 2 weeks of assigned treatment
  Protein, if present, measured in urine in complete urinalysis
Protein in urine | 4 weeks of assigned treatment
  Protein, if present, measured in urine in complete urinalysis
Glucose in urine | baseline
  Glucose, if present, measured in urine in complete urinalysis
Glucose in urine | 2 weeks of assigned treatment
  Glucose, if present, measured in urine in complete urinalysis
Glucose in urine | 4 weeks of assigned treatment
  Glucose, if present, measured in urine in complete urinalysis
Ketones in urine | baseline
  Ketones, if present, measured in urine in complete urinalysis
Ketones in urine | 2 weeks of assigned treatment
  Ketones, if present, measured in urine in complete urinalysis
Ketones in urine | 4 weeks of assigned treatment
  Ketones, if present, measured in urine in complete urinalysis
Occult blood in urine | baseline
  Occult blood, if present, measured in urine in complete urinalysis
Occult blood in urine | 2 weeks of assigned treatment
  Occult blood, if present, measured in urine in complete urinalysis
Occult blood in urine | 4 weeks of assigned treatment
  Occult blood, if present, measured in urine in complete urinalysis
White blood cell esterase in urine | baseline
  White blood cell esterase, if present, measured in urine
White blood cell esterase in urine | 2 weeks of assigned treatment
  White blood cell esterase, if present, measured in urine
White blood cell esterase in urine | 4 weeks of assigned treatment
  White blood cell esterase, if present, measured in urine
Urine nitrite | baseline
  nitrite, if present, measured in urine
Urine nitrite | 2 weeks of assigned treatment
  nitrite, if present, measured in urine
Urine nitrite | 4 weeks of assigned treatment
  nitrite, if present, measured in urine
bilirubin in urine | baseline
  bilirubin, if present, measured in urine
bilirubin in urine | 2 weeks of assigned treatment
  bilirubin, if present, measured in urine
bilirubin in urine | 4 weeks of assigned treatment
  bilirubin, if present, measured in urine
urobilinogen in urine | baseline
  urobilinogen in urine measured in urinalysis as mg/dL
urobilinogen in urine | 2 weeks of assigned treatment
  urobilinogen in urine measured in urinalysis as mg/dL
urobilinogen in urine | 4 weeks of assigned treatment
  urobilinogen in urine measured in urinalysis as mg/dL
Heart Rate | baseline
  Heart Rate measured using an automated blood pressure machine
Heart Rate | 2 weeks of assigned treatment
  Heart rate measured using an automated blood pressure machine
Heart Rate | 4 weeks of assigned treatment
  Heart rate measured using an automated blood pressure machine
Blood Pressure | baseline
  Systolic and Diastolic blood pressure measured using an automated blood pressure machine
Blood Pressure | 2 weeks of assigned treatment
  Systolic and Diastolic blood pressure measured using an automated blood pressure machine
Blood Pressure | 4 weeks of assigned treatment
  Systolic and Diastolic blood pressure measured using an automated blood pressure machine
Product Tolerability questionnaire (gastrointestinal) | baseline
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the past two weeks from 0 (None) to 10 (severe)
Product Tolerability questionnaire (gastrointestinal) | 2 weeks of assigned treatment
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the past two weeks from 0 (None) to 10 (severe)
Product Tolerability questionnaire (gastrointestinal) | 4 weeks of assigned treatment
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the past two weeks from 0 (None) to 10 (severe)
Product Tolerability questionnaire (consumption) | baseline
  Questionnaire that can be scored 1-5 (1 bad quality to 5 good quality): answers of strongly agree, agree, neutral, disagree, and strongly agree for tastes pleasant, easy to drink, easy on stomach, would purchase, dissolves easily, too gritty, too sticky and excessively, mildly too much, optimal, mildly too little, and extremely lacking for sweet, sour, salty, bitter. Final question on after taste with answers of pleasant, ok, no taste, unpleasant, extremely unpleasant.
Product Tolerability questionnaire (consumption) | 2 weeks of assigned treatment
  Questionnaire that can be scored 1-5 (1 bad quality to 5 good quality): with answers of strongly agree, agree, neutral, disagree, and strongly agree for tastes pleasant, easy to drink, easy on stomach, would purchase, dissolves easily, too gritty, too sticky and excessively, mildly too much, optimal, mildly too little, and extremely lacking for sweet, sour, salty, bitter. Final question on after taste with answers of pleasant, ok, no taste, unpleasant, extremely unpleasant.
Product Tolerability questionnaire (consumption) | 4 weeks of assigned treatment visit
  Questionnaire that can be scored 1-5 (1 bad quality to 5 good quality): with answers of strongly agree, agree, neutral, disagree, and strongly agree for tastes pleasant, easy to drink, easy on stomach, would purchase, dissolves easily, too gritty, too sticky and excessively, mildly too much, optimal, mildly too little, and extremely lacking for sweet, sour, salty, bitter. Final question on after taste with answers of pleasant, ok, no taste, unpleasant, extremely unpleasant.
tolerability questionnaire | 3 days before baseline visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 3 days before baseline visit
  A list of all food and drink consumed that day
tolerability questionnaire | 2 days before baseline visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 2 days before baseline visit
  A list of all food and drink consumed that day
tolerability questionnaire | 1 day before baseline visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 1 day before baseline visit
  A list of all food and drink consumed that day
tolerability questionnaire | 3 days before 2 week visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 3 days before 2 week visit
  A list of all food and drink consumed that day
Daily food diary | 2 days before 2 week visit
  A list of all food and drink consumed that day
tolerability questionnaire | 2 days before 2 week visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
tolerability questionnaire | 1 day before 2 week visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 1 day before 2 week visit
  A list of all food and drink consumed that day
tolerability questionnaire | 3 days before 4 week visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 3 days before 4 week visit
  A list of all food and drink consumed that day
tolerability questionnaire | 2 days before 4 week visit
  A list of all food and drink consumed that day along with a Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 2 days before 4 week visit
  A list of all food and drink consumed that day
tolerability questionnaire | 1 day before 4 week visit
  Visual analog scale used to assess gastrointestinal issues (bloating, constipation, diarrhea, frequent urination, gas, nausea, stomach fullness, abdominal pain/cramping) over the day (None) to 10 (severe)
Daily food diary | 1 day before 4 week visit
  A list of all food and drink consumed that day

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States